CLINICAL TRIAL: NCT07210164
Title: Prehabilitation With Exercise and Immunonutrition (Ocoxin®) in the Perioperative Management of Gynecologic Malignancies Under ERAS Protocol.
Brief Title: Pre-habilitation Within ERAS Protocol for Gynecologic Oncology Surgery: The Pre_ERAS Study
Acronym: Pre_ERAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Catalysis SL (Industry)
Responsible Party: Principal Investigator, Panagiotis Tzitzis, MD,MSc, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 337/2025, 18.09.2025
Record Dates: First submitted 2025-09-18; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: ERAS; Compliance; Quality of Life (QOL); Excercise; Immunonutrition; Post Operative Pain; Laparotomy Patients; Surgical Complication; Gynaecological Malignancies; Gynaecologic Cancer; Gynaecological Oncology
Keywords: Prehabilitation; ERAS; Gynecologic Cancers; Immunonutrition
MeSH Terms: conditions — Patient Compliance; Pain, Postoperative | interventions — Ocoxin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation group (Experimental): This group undergo a structured preoperative self-guided exercise protocol (consisting of mild physical activity with a defined exercise program, respiratory exercise, muscle strengthening), immunonutrition (Ocoxin©) and usual clinical practice (stopping alcohol, regulating anemia and glucose levels). During the period of hospitalatization adhere to the 21-point ERAS protocol .
  Interventions: Dietary Supplement: Ocoxin; Procedure: Structured self-guided exercise
- Control group (No Intervention): This group follow the usual clinical practice (stopping alcohol, regulating anemia and glucose levels). During the period of hospitalatization adhere to the 21-point ERAS protocol .

INTERVENTIONS:
Dietary Supplement: Ocoxin — Food Supplement based on Amino Acids, Plants, Vitamins and Minerals. Composition: Maltodextrin, L-Arginine, L-Cysteine, Microcrystalline cellulose, Talcum, Vitamin C (L-ascorbic acid), Zinc sulfate, Green Tea Extract (Camellia sinensis (L.) Kuntze), Manganese sulphate, Extracto de Canela (Cinnamomum verum J. Presl.), Vitamin B6 (pyridoxine hydrochloride).
  Ocoxin utilizes Catalysis' Molecular Activation Technology (MAT) to enhance the biological activity of its natural antioxidant ingredients, such as green tea polyphenols (EGCG), to increase their antitumoral and immunomodulatory effects. This patented technology is applied to boost the efficacy of compounds within Ocoxin, such as EGCG, enabling them to exert more potent effects on cancer cells by inducing apoptosis, inhibiting tumor growth and metastasis, and supporting the body's immune response.
  Arms: Prehabilitation group
Procedure: Structured self-guided exercise — The patient exercises in a structured manner with the help of a relevant interactive form/guide and simple aids (e.g. chair, step, water bottle, broomstick) by performing six categories of exercises: 1. Breathing exercises, 2. Pelvic floor exercises-pelvic mobility, 3. Upper trunk exercises, 4. Lower trunk exercises, 5. Aerobic exercises, 6. Stretching exercises, at a predetermined pace (number of repetitions) of each exercise and a limit of not exceeding the value 5-6 on the ten-point modified Borg fatigue scale. The intern records her activity on a form-"exercise log". The recommendation is the maximum implementation of the exercise program but in any case not less than 3 times a week.
  Arms: Prehabilitation group

SUMMARY:
ERAS (Enhanced Recovery After Surgery) protocols are step-by-step care plans that help patients recover faster after surgery. They focus on keeping the body's normal functions, lowering stress from surgery, and supporting a quicker recovery. In gynecologic cancer surgeries, ERAS has been shown to help patients do better, have fewer problems, and leave the hospital sooner.

A prehabilitation program, in combination with ERAS protocols, aims to optimize patients' physical and psychological condition prior to surgery for gynecological cancers. Interventions may include tailored exercise, nutritional support, respiratory training, and psychological preparation. By enhancing baseline fitness and resilience, prehabilitation improves the body's ability to tolerate surgical stress, reduces complications, and facilitates a faster, smoother recovery within the ERAS framework.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the impact of multifactorial preoperative empowerment (pre-habilitation protocol) on patients with gynecological cancer who undergo oncological surgery. The objective of this study is to demonstrate whether the implementation of pre-habilitation program empowerment as opposed to its non-implementation leads to an improvement in quality of life, a reduction in days of hospitalization, a reduction in immediate (up to discharge) and long term (up to 40th post-surgery day) postoperative complications (as measured with the Clavien Dindo system), a reduction in hospital readmission rates, and postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Type of gynecological malignancy: endometrial cancer, ovarian cancer, cervical cancer, treated with laparotomy after the decision of the gynecological-oncology unit (positive opinion of the Multidisciplinary Tumor Board - MDT)
* Patient age: 18 to 85 years
* General condition of the patient: ASA score I-III
* Consent to implement the accelerated recovery protocol - Enhanced recovery after surgery (ERAS)
* Sufficient understanding of the Greek language
* Provision of signed, after thorough information, consent to participate in the study

Exclusion Criteria:

* Women with performance status: ECOG >2 and ASA score >III
* Women who have not been informed and have given written consent

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-30 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative morbidity | Up to the 30th post operative day
  Systematic recording of complications based on the Clavien Dindo system, during hospitalization and in the immediate postoperative period (up to the 30th postoperative day).
Duration of hospitalization | Until the patient discharged (assessed up to 4 days)
  The discharge day is defined as the postoperative day on which the following criteria are met in their entirety: 1. adequate mobilization, 2. tolerance of solid foods and adequate oral water intake, 3. adequate analgesia only with oral analgesics, 4. mobilization of intestinal function / flatus, 5. Absence of Clavien Dindo >II complication.
General Quality of Life (QoL) | Up to the time of discharge (assessed up to 4 days)
  Use of metric tools: structured and weighted questionnaires in Greek language EORTC QLQ-C30 (version 3.0) (general quality of life).
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items.
  Each of the multi-item scales includes a different set of items - no item occurs in more than one scale.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.

SECONDARY OUTCOMES:
Time interval between the onset of adjuvant anti-neoplastic therapy | Up to 120 days after surgery
  The number of days between the day of surgery and the start of adjuvant therapy (includes systemic chemotherapy/immunotherapy, external radiation, brachytherapy).
Hospital readmission at 90 days | Up to the 90th postoperative day
  Any admission to a nursing facility up to the 90th postoperative day.
Cachexia | Up to the time of discharge (assessed up to 5 days)
  Assessments using unique measurements EORTC QLQ-CAX24 (cachexia). The Cancer Cachexia Module is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-CAX24 incorporates five multi-item scales to assess food aversion, eating and weight-loss worry, eating difficulties, loss of control, and physical decline. In addition, four single items assess dry mouth, indigestion/heartburn, forcing self to eat and inadequate information.
  All of the scales and single-item measures range in score from 0 to 100. A high score for the symptom scales represents a high level of symptomatology or problems.
Sexual Health | Up to the time of discharge (assessed up to 4 days)
  The EORTC Quality of Life Questionnaire Sexual Health (SH-22) is a stand-alone questionnaire, but can also be used as a supplementary questionnaire to be employed in conjunction with the QLQ-C30. The SH-22 incorporates 2 multi-item scales to assess Sexual satisfaction and Sexual pain. In addition, 11 single items assess sexual activity and cover treatment-related and partner-related questions, general questions of sexual health and 4 gender specific questions.
  Interpretation: All of the Multi-item scales and Single-item measures range in score from 0 to 100. A high score represents a high level of symptomatology or problems.
  Reporting: The two multi-item scales have a different number of items depending on whether the patient had or does not have a partner, and has or does not have sexual activity. It is advised to always report how many items were used to calculate each scale; and which ones. This will allow comparison between different subgroups of patients.
Quality of Life in ovarian cancer | Up to the time of discharge (assessed up to 4 days)
  The Ovarian Cancer Module (QLQ-OV28) is a supplementary questionnaire module to be employed in conjunction with the QLQ-C30. The QLQ-OV28 incorporates seven multi-item scales to assess body image, sexuality, attitude to disease or treatment, abdominal or gastro-intestinal symptoms, peripheral neuropathy, hormonal or menopausal symptoms and other chemotherapy side-effects.
  The scoring approach for the QLQ-OV28 is identical in principle to that for the [function and/or symptom scales / single items] of the QLQ-C30.
  Interpretation: All of the scales and single-item measures range in score from 0 to 100. A high score for the [functional scales and/or single items] represents a high level of functioning, whereas a high score for the [symptom scales and/or single items] represents a high level of symptomatology or problems.
Quality of Life in endometrial cancer | Up to the time of discharge (assessed up to 4 days)
  The Endometrial Cancer Module (QLQ-EN24) is a supplementary questionnaire module designed for patients with all stages of endometrial cancer and should always be employed in conjunction with the QLQ-C30. The QLQ-EN24 incorporates 5 multi-item scales to assess lymphoedema, urological symptoms, gastrointestinal symptoms, body image and sexual/vaginal problems. In addition, 8 single items assess pain in back and pelvis, tingling/numbness, muscular pain, hair loss, taste change, sexual interest, sexual activity and sexual enjoyment.
  The scoring approach for the QLQ-EN24 is identical in principle to that for the symptom scales/single-items of the QLQ-C30.
  Interpretation:
  All of the scales and single-item measures range in score from 0 to 100. A high score for the functional items represents a high level of functioning, whereas a high score for the symptom scales and single-items represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios C. Tsolakidis, MD, PhD, Study Chair — Professor of Obstetrics - Gynaecology, Aristotel University of Thessaloniki; Panagiotis M. Tzitzis, MD, MSc, Principal Investigator — PhD (c) 1st Department of Obstetrics - Gynaecology Aristotel University of Thessaloniki
Locations (1):
- General Hospital of Papageorgiou, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for pre- and intra-operative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part I. Gynecol Oncol. 2016 Feb;140(2):313-22. doi: 10.1016/j.ygyno.2015.11.015. Epub 2015 Nov 18. No abstract available. PMID 26603969
- [Background] Miralpeix E, Mancebo G, Gayete S, Corcoy M, Sole-Sedeno JM. Role and impact of multimodal prehabilitation for gynecologic oncology patients in an Enhanced Recovery After Surgery (ERAS) program. Int J Gynecol Cancer. 2019 Oct;29(8):1235-1243. doi: 10.1136/ijgc-2019-000597. Epub 2019 Aug 30. PMID 31473663
- [Background] Nelson G, Altman AD, Nick A, Meyer LA, Ramirez PT, Achtari C, Antrobus J, Huang J, Scott M, Wijk L, Acheson N, Ljungqvist O, Dowdy SC. Guidelines for postoperative care in gynecologic/oncology surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations--Part II. Gynecol Oncol. 2016 Feb;140(2):323-32. doi: 10.1016/j.ygyno.2015.12.019. Epub 2016 Jan 3. No abstract available. PMID 26757238
- [Background] Hubner M, Kusamura S, Villeneuve L, Al-Niaimi A, Alyami M, Balonov K, Bell J, Bristow R, Guiral DC, Fagotti A, Falcao LFR, Glehen O, Lambert L, Mack L, Muenster T, Piso P, Pocard M, Rau B, Sgarbura O, Somashekhar SP, Wadhwa A, Altman A, Fawcett W, Veerapong J, Nelson G. Guidelines for Perioperative Care in Cytoreductive Surgery (CRS) with or without hyperthermic IntraPEritoneal chemotherapy (HIPEC): Enhanced Recovery After Surgery (ERAS(R)) Society Recommendations - Part II: Postoperative management and special considerations. Eur J Surg Oncol. 2020 Dec;46(12):2311-2323. doi: 10.1016/j.ejso.2020.08.006. Epub 2020 Aug 13. PMID 32826114
- [Background] Bisch SP, Jago CA, Kalogera E, Ganshorn H, Meyer LA, Ramirez PT, Dowdy SC, Nelson G. Outcomes of enhanced recovery after surgery (ERAS) in gynecologic oncology - A systematic review and meta-analysis. Gynecol Oncol. 2021 Apr;161(1):46-55. doi: 10.1016/j.ygyno.2020.12.035. Epub 2020 Dec 30. PMID 33388155
- [Background] Miralpeix E, Fabrego B, Rodriguez-Cosmen C, Sole-Sedeno JM, Gayete S, Jara-Bogunya D, Corcoy M, Mancebo G. Prehabilitation in an ERAS program for endometrial cancer patients: impact on post-operative recovery. Int J Gynecol Cancer. 2023 Apr 3;33(4):528-533. doi: 10.1136/ijgc-2022-004130. PMID 36898697
- [Background] Ferrero A, Vassallo D, Geuna M, Fuso L, Villa M, Badellino E, Barboni M, Coata P, Santoro N, Delgado Bolton RC, Biglia N. Immunonutrition in ovarian cancer: clinical and immunological impact? J Gynecol Oncol. 2022 Nov;33(6):e77. doi: 10.3802/jgo.2022.33.e77. Epub 2022 Aug 12. PMID 36047379
- [Background] Prieto I, Montemuino S, Luna J, de Torres MV, Amaya E. The role of immunonutritional support in cancer treatment: Current evidence. Clin Nutr. 2017 Dec;36(6):1457-1464. doi: 10.1016/j.clnu.2016.11.015. Epub 2016 Nov 24. PMID 27931879
- [Background] Nelson G, Bakkum-Gamez J, Kalogera E, Glaser G, Altman A, Meyer LA, Taylor JS, Iniesta M, Lasala J, Mena G, Scott M, Gillis C, Elias K, Wijk L, Huang J, Nygren J, Ljungqvist O, Ramirez PT, Dowdy SC. Guidelines for perioperative care in gynecologic/oncology: Enhanced Recovery After Surgery (ERAS) Society recommendations-2019 update. Int J Gynecol Cancer. 2019 May;29(4):651-668. doi: 10.1136/ijgc-2019-000356. Epub 2019 Mar 15. PMID 30877144
- [Background] Nelson G, Fotopoulou C, Taylor J, Glaser G, Bakkum-Gamez J, Meyer LA, Stone R, Mena G, Elias KM, Altman AD, Bisch SP, Ramirez PT, Dowdy SC. Enhanced recovery after surgery (ERAS(R)) society guidelines for gynecologic oncology: Addressing implementation challenges - 2023 update. Gynecol Oncol. 2023 Jun;173:58-67. doi: 10.1016/j.ygyno.2023.04.009. Epub 2023 Apr 21. PMID 37086524
- [Background] Bisch S, Nelson G, Altman A. Impact of Nutrition on Enhanced Recovery After Surgery (ERAS) in Gynecologic Oncology. Nutrients. 2019 May 16;11(5):1088. doi: 10.3390/nu11051088. PMID 31100877
- [Background] Arends J, Bachmann P, Baracos V, Barthelemy N, Bertz H, Bozzetti F, Fearon K, Hutterer E, Isenring E, Kaasa S, Krznaric Z, Laird B, Larsson M, Laviano A, Muhlebach S, Muscaritoli M, Oldervoll L, Ravasco P, Solheim T, Strasser F, de van der Schueren M, Preiser JC. ESPEN guidelines on nutrition in cancer patients. Clin Nutr. 2017 Feb;36(1):11-48. doi: 10.1016/j.clnu.2016.07.015. Epub 2016 Aug 6. PMID 27637832
- [Background] Diaz-Feijoo B, Agusti-Garcia N, Sebio R, Lopez-Hernandez A, Siso M, Glickman A, Carreras-Dieguez N, Fuste P, Marina T, Martinez-Egea J, Aguilera L, Perdomo J, Pelaez A, Lopez-Baamonde M, Navarro-Ripoll R, Gimeno E, Campero B, Torne A, Martinez-Palli G, Arguis MJ. Feasibility of a Multimodal Prehabilitation Programme in Patients Undergoing Cytoreductive Surgery for Advanced Ovarian Cancer: A Pilot Study. Cancers (Basel). 2022 Mar 23;14(7):1635. doi: 10.3390/cancers14071635. PMID 35406407
- [Background] Inci MG, Sehouli J, Schnura E, Lee M, Roll S, Reinhold T, Klews J, Kaufner L, Niggemann P, Groeben H, Toelkes J, Reisshauer A, Liebl M, Daehnert E, Zimmermann M, Knappe-Drzikova B, Rolker S, Nunier B, Algharably E, Pirmorady Sehouli A, Zwantleitner L, Krull A, Heitz F, Ataseven B, Chekerov R, Harter P, Schneider S. The KORE-INNOVATION trial, a prospective controlled multi-site clinical study to implement and assess the effects of an innovative peri-operative care pathway for patients with ovarian cancer: rationale, methods and trial design. Int J Gynecol Cancer. 2023 Aug 7;33(8):1304-1309. doi: 10.1136/ijgc-2023-004531. PMID 37208019